CLINICAL TRIAL: NCT04756635
Title: Effects of Short- Term Intermittent Fasting on Neuromuscular Performance, Aerobic and Anaerobic Capacity
Brief Title: Effects of Short- Term Intermittent Fasting Aerobic and Anaerobic Capacity
Acronym: Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Principal Investigator, Joana Correia, Principal Investigator, Faculdade de Motricidade Humana
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: joana_correia
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Healthy Males; Men
Keywords: Intermittent fasting; neuromuscular performance; aerobic capacity; anaerobic capacity
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Measures taken before and after the defined IF periods. Two groups of participants will be included in this project: 1) resistance trained group (tested for neuromuscular function, anaerobic capacity and body composition); 2) endurance trained group (tested for aerobic and anaerobic capacity and body composition). Experimental condition: pre- and post-4 weeks of IF. Measurements will be taken during the morning period (between 07:00 and 11:00 am) in the fasted state. Neuromuscular function and anaerobic capacity will be assessed on separate days (with at least a 48- hour interval) to ensure full recovery.
  Interventions: Other: Experimental Group
- Control Group (Other): Participants of each group serving as their own controls. Control condition: pre- and post4 weeks of normal diet. Measurements will be taken during the morning period (between 07:00 and 11:00 am) in the fasted state. Neuromuscular function and anaerobic capacity will be assessed on separate days (with at least a 48-hour interval) to ensure full recovery.
  Interventions: Other: Experimental Group

INTERVENTIONS:
Other: Experimental Group — This 3-year project will include two groups of participants: 1) young men accustomed to resistance training (study #1) and 2) young men accustomed to endurance training (study #2). Inclusion will be limited to healthy participants (i.e. nonsmokers, normotensive with systolic and diastolic values <135/85 mmHg, non-obese, non-medicated, and free of any known disease as assessed by medical history) (Pickering, Hall et al. 2005). Month 1-3 will focus on literature review and month 4 to 8 will address experimental settings preparation and selection of participants to include in each study. Testing and data collection will be scheduled for months 9-14 and 13-18 (study # 1 and 2 related testing, respectively). Data processing, analysis and presentation will occur from month 21 to 33. All participants will read and sign an informed consent document with the description of the testing procedures. The Faculty's ethical committee will be asked to approve this document before testing.
  Other Names: Aerobic capacity; Anaerobic capacity; Neuromuscular performance

SUMMARY:
The therapeutic use of caloric restriction and intermittent fasting (IF) protocols improves life span and health related quality of life. The effects of fasting protocols on athletic performance and training adaptations have been primarily studied in athletes undergoing the Ramadan IF protocol or in athletes willing to decrease body fat, while maintaining or increasing lean body mass. Data from these studies are somewhat conflicting and unclear. Moreover, the effects of IF on muscular strength, as well as in aerobic and anaerobic capacity remain largely unknown. Anecdotal evidence from experienced participants in strength, power and endurance training or sports, indicates an increased ability to acutely display higher levels of work capacity in the fasted vs. fed state. The goal of this project is to determine the effects of 4 wks of IF on neuromuscular performance, aerobic and anaerobic capacity of well-trained young adults.

DETAILED DESCRIPTION:
This 3-year project will include two groups of participants: 1) young men accustomed to resistance training (study #1) and 2) young men accustomed to endurance training (study #2). Inclusion will be limited to healthy participants (i.e. nonsmokers, normotensive with systolic and diastolic values <135/85 mmHg, non-obese, non-medicated, and free of any known disease as assessed by medical history) (Pickering, Hall et al. 2005). Month 1-3 will focus on literature review and month 4 to 8 will address experimental settings preparation and selection of participants to include in each study. Testing and data collection will be scheduled for months 9-14 and 13-18 (study # 1 and 2 related testing, respectively). Data processing, analysis and presentation will occur from month 21 to 33. All participants will read and sign an informed consent document with the description of the testing procedures. The Faculty's ethical committee will be asked to approve this document before testing. All studies will follow a randomized crossover design, with measures taken before and after the defined IF periods and participants of each group serving as their own controls. Two groups of participants will be included in this project: 1) group #1: resistance trained group (tested for neuromuscular function, anaerobic capacity and body composition); 2) group #2: endurance trained group (tested for aerobic and anaerobic capacity and body composition). In a randomized, counterbalanced manner, all participants will be tested in two different conditions: control condition (pre- and post4 wks of normal diet) vs. experimental condition (pre- and post-4 wks of IF). A 2-wk washout period will separate both conditions. Measurements will be taken during the morning period (between 07:00 and 11:00 am) in the fasted state. Neuromuscular function and anaerobic capacity will be assessed on separate days (with at least a 48- hour interval) to ensure full recovery.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion will be limited to young, healthy men with aged 20- 30 years. All participants will exhibit > 3 years of continued experience and current participation in strength and power sports/training (training frequency of at least 3 times/wk). As importantly, the following criteria will also be determinant for inclusion: 1) bench press one-repetition maximum/bodyweight ratio > 1.26 (i.e. above the 80 percentile for 20 to 29-year-old males) (ACSM 2013) and 2) leg press one-repetition maximum /bodyweight ratio > 2.08 (i.e. above the 80 percentile for 20 to 29-year-old males) (ACSM 2013). Finally, for inclusion, all participants will have to follow the nutritional and training recommendations at pre-testing time point.
* For study 2, as for study 1, Inclusion will be limited to young, healthy men with aged 20- 30 yrs. All participants will exhibit > 3 yrs of continued experience and current participation in endurance based sports/training (training frequency of at least 3 times/wk). We will only include participants with VO2peak values > 49 mL.kg-1.min-1(i.e. above the 80 percentile for 20 to 29-year-old males) (ACSM 2013). Finally, for inclusion, all participants will have to follow the nutritional and training recommendations at pre-testing time point.

Exclusion Criteria:

* All participants who do not meet the inclusion criteria mentioned above.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2023-02-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Performance at 4 weeks | 4weeks (experiemental) + 4weeks (control)
  Neuromuscular performance, aerobic and anaerobic capacity

SECONDARY OUTCOMES:
Change from Baseline Body Composition at 4 weeks | 4weeks (experiemental) + 4weeks (control)
  Fat Free Mass (kilograms), Fat Mass (kilograms), Body Mass Index (kg/m^2), Body Weight (kilograms)

CONTACTS AND LOCATIONS:
Overall Officials: Joana M. Correia, Master, Principal Investigator — Faculdade de Motricidade Humana
Locations (1):
- Joana Correia, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Public articles with no reference to participants
Supporting Information: Study Protocol, CSR
Time Frame: The data will be stored in an SPSS and excel database, on the server of the Faculty of Human Motricity assigned to the Motor Behavior Laboratory. Paper-based documents will be destroyed after the data processing matrix is built.
Access Criteria: Public articles with no reference to participants

REFERENCES:
- [Derived] Correia JM, Pezarat-Correia P, Minderico C, Infante J, Mendonca GV. Effects of Time-Restricted Eating on Aerobic Capacity, Body Composition, and Markers of Metabolic Health in Healthy Male Recreational Runners: A Randomized Crossover Trial. J Acad Nutr Diet. 2024 Aug;124(8):1041-1050. doi: 10.1016/j.jand.2024.01.005. Epub 2024 Jan 17. PMID 38242204